CLINICAL TRIAL: NCT01614041
Title: Tandospirone Citrate in the Treatment of Patients With Generalized Anxiety Disorder: a Multi-center, Randomized, Usual Dose-controlled Trial
Brief Title: Tandospirone Citrate in the Treatment of Patients With Generalized Anxiety Disorder
Acronym: TACGAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSPC-SED-1101
Record Dates: First submitted 2011-11-11; First posted 2012-06-07 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Patient randomized to control group is administrated with usual dose of tandospirone treatment, 30 mg/day
  Interventions: Drug: Usual dose treatment of Tandospirone
- Study Group (Experimental): Comparative high dose of tandospirone treatment, 60 mg/day
  Interventions: Drug: Comparative high dose of tandospirone treatment

INTERVENTIONS:
Drug: Usual dose treatment of Tandospirone — Usual dose treatment of Tandospirone, oral, 30 mg/day
  Arms: Control Group
Drug: Comparative high dose of tandospirone treatment — Comparative high dose of tandospirone treatment, oral, 60 mg/day
  Arms: Study Group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of comparative high dose Tandospirone Citrate in the treatment of patients with generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Male or female
* Diagnosed with GAD according to DSM-IV
* HAMA score≥17
* Provide with written informed consent
* Agree to be washed-out for two weeks if receiving SSRI, SNRI or NASA.

Exclusion Criteria:

* Serious suicidal tendency
* The score of the sixth item of HAMA ≥3
* The score of HAMD ≥21
* Pregnant or lactating women
* History of allergic or hypersensitivity to tandospirone
* Serious or unstable cardiac, renal, neurologic, cerebrovascular, metabolic, or pulmonary disease
* Secondary anxiety disorders
* Drug or alcohol dependence within 1 year
* Patients currently taking benzodiazepine drugs
* Drivers and dangerous machine operators
* Participated in other clinical studies in the last 30 days
* Patients with clinically significant ECG or laboratory abnormalities
* Patients with a history of epilepsy
* Patients with abnormal TSH concentration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2012-01-10 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients whose Hamilton Anxiety Scale (HAMA) score change downwards ≥ 50% from baseline to 6 weeks treatment | 6 weeks
  HAMA score changes downwards ≥ 50% indicate significant improvement; HAMA score changes downwards ≥ 75% indicate remission

SECONDARY OUTCOMES:
HAMA score changes from baseline to 6 weeks treatment | 6 weeks
  Scores 14-21 indicate mild anxiety; scores 21-29 indicate moderate anxiety; scores over 29 indicate severe anxiety
Percentage of patients whose HAMA score ≤ 7 after 6 weeks treatment | 6 weeks
  Scores ≤ 7 indicate non-anxious
HAMA factor score changes after treatment | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wenyuan Wu, MD, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Shanghai, China

REFERENCES:
- [Derived] Fu Y, Ji JL, Shi SX, Zhang HY, Lin GZ, Zhang YL, Li X, Wu WY. Early outcomes, associated factors and predictive values of clinical outcomes of tandospirone in generalized anxiety disorder: a post-hoc analysis of a randomized, controlled, multicenter clinical trial. Curr Med Res Opin. 2023 Apr;39(4):597-603. doi: 10.1080/03007995.2023.2175998. Epub 2023 Feb 26. PMID 36842964
- [Derived] Li Q, Zhang H, Lin G, Shi S, Zhang Y, Ji J, Yang L, Yao J, Wu W. Relative Safety and Efficacy of Two Doses of Tandospirone Citrate for Generalized Anxiety Disorder: A Multicenter Randomized Controlled Trial. Neuropsychiatr Dis Treat. 2022 Aug 8;18:1653-1664. doi: 10.2147/NDT.S366048. eCollection 2022. PMID 35968511